CLINICAL TRIAL: NCT05547035
Title: Prospective, Multicenter Non-randomised, Open-label Study Evaluating the Correlation Between Physiological Data Measured by a Portable Sensor and Psychometric Assessment
Brief Title: Identification of Physiological Data by a Wearable Monitor in Subjects Suffering From Major Depression Disorders
Acronym: MYND104
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Digital For Mental Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-A00595-48; 2017-A00595-48 (Other: French Competent Authority(ANSM) reference number)
Record Dates: First submitted 2022-07-01; First posted 2022-09-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable monitor collected phydiological measurements (Experimental): This is a single arm study with a wearable monitor that collects physiological measures (falling in the categories physical activity, heart rate, heart rate variability, breathing rate and sleep) 24/7 in ambulatory.
  Interventions: Behavioral: Patient follow-up of depression

INTERVENTIONS:
Behavioral: Patient follow-up of depression — All patients who agree to participate in the study are diagnosed by their GP/Psychiatrist with a diagnostic assessment instrument called DSM-5. Participants visit their GPs/Psychiatrists at baseline, month 1, month 2, month 3, month 4, month 5 and month 6. At each visit, the GPs/Psychiatrists:
  * assess the depression severity by using MADRS scale
  * assess the severity of illness at time of assessment compared with start of treatment by using CGI-S measures
  * the patient complete the self-administered questionnaire of HAD scale that measures the symptoms of anxiety and depression.

SUMMARY:
To evaluate, over a period of six months, the links between physiological data collected such as electrodermal activity (or Galvanic Skin Response), motor activity measured by accelerometer, heartbeat measured by photoplestimograph and the clinical evaluation performed by the physician, in patients suffering from major depression disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patient able to give written informed consent, - Presenting a major depressive episode defined according to DSM V criteria, - Presenting a MADRS score ≥ 20 - Able to understand all study procedures and follow-up

Exclusion Criteria:

* - Inability to wear the wearable monitor for the duration of the study (6 months)
* Patient with a severe medical condition at the discretion of the investigator (neurological, rheumatological, etc.)
* Resistant depression
* Chronic depression, dysthymia
* Depression with psychotic features not congruent with mood, schizophrenia disorder
* Depression with catatonic features
* Substance use disorder in the last 6 months
* Extreme sports during the conduct of the study
* Pre-existing skin infection at the wearable monitor site
* Pregnant or lactating woman
* Participation in another drug or medical device study
* Inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in MADRS ( Montgomery-Asberg Depression Rating Scale) total score with physiological measurements. | Baseline, Month1, Month 2, Month 3, Month 4, Month 5, Month 6
  * Change in central rater Montgomery-Asberg Depression Rating Scale (MADRS) total score and comparison with changes in physiological measurements such as activity, emotional arousal, heart rate, heart rate variability, breathing rate and sleep.
  * The Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is rated on a scale of 0 to 6, with differing descriptors for each item. These individual item scores are added together to form a total score, which can range between 0 (low severity of depressive symptoms) and 60 points (high severity of depressive symptoms), higher score indicating poorer health outcomes. The MADRS provides a measure of the overall level of depression.
Comparison of change in HAD (Hospital Anxiety and Depression) total score with physiological measurements. | Baseline, Month1, Month 2, Month 3, Month 4, Month 5, Month 6
  * Change in Hospital Anxiety and Depression total score and comparison with changes in physiological measurements such as activity, emotional arousal, heart rate, heart rate variability, breathing rate and sleep.
  * The Hospital Anxiety and Depression Scale used for measuring anxiety Scored on a scale of 0-21 (higher score more anxiety) and for measuring depression Scored on a scale of 0-21 (higher score more depression).
Comparison of change in CGI (Clinical Global Impression) scale with physiological measurements. | Baseline, Month1, Month 2, Month 3, Month 4, Month 5, Month 6
  * Change in CGI scale and comparison with changes in physiological measurements such as activity, emotional arousal, heart rate, heart rate variability, breathing rate and sleep.
  * The Clinical Global Impression Scale (CGI-s), is a widely administered clinician rated scale that assesses the subject overall illness severity and the degree of improvement from the initial assessment. Illness severity is rated on a 1-7 scale where 1 corresponds to "Normal, Not at All Ill", 2 is "Borderline Mentally Ill", the anchor for 3 is "Mildly Ill", the anchor for 4 is "Moderately Ill", 5 is "Markedly Ill", 6 is "Severely Ill", and 7 is "Among the Most Extremely Ill Patients".The degree of improvement is rated on a 1-7 scale where 1 corresponds to "Very Much Improved", 2 is "Much Improved", the anchor for 3 is "Minimally Improved", the anchor for 4 is "No Change", 5 is "Minimally Worse", 6 is "Much Worse", and 7 is "Very Much Worse".

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - 135 rue Nestor Longue Epee, Bersée
  - 203 rue de la Motte, Bersée
  - APPT 22 Residence les Tilleuls, Dax
  - 2 boulevard Winston Churchill, Dijon
  - Clinique Lyon Lumiere, Meyzieu
  - 22 rue Jacques Boutrolles, Mont-Saint-Aignan
  - 19 rue de la Liberté, Nice
  - 119 rue de la Pompe, Paris
  - 91 rue Caulaincpurt, Paris
  - 145 avenue des Minimes, Toulouse